CLINICAL TRIAL: NCT02595866
Title: Phase I Study of MK-3475 (Pembrolizumab) in Patients With Human Immunodeficiency Virus (HIV) and Relapsed/Refractory or Disseminated Malignant Neoplasm
Brief Title: Testing the Addition of an Experimental Medication MK-3475 (Pembrolizumab) to Usual Anti-Retroviral Medications in Patients With HIV and Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01906; NCI-2015-01906 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); s16-01365; CITN-12 (Other: Cancer Immunotherapy Trials Network); CITN-12 (Other: CTEP); P30CA015704 (NIH); U01CA154967 (NIH)
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Results first posted 2024-07-16 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-05

CONDITIONS: AIDS-Related Non-Hodgkin Lymphoma; Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Hepatocellular Carcinoma; HIV Infection; Kaposi Sarcoma; Locally Advanced Lung Non-Small Cell Carcinoma; Locally Advanced Malignant Solid Neoplasm; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Malignant Solid Neoplasm; Metastatic Melanoma; Non-Hodgkin Lymphoma; Recurrent Classic Hodgkin Lymphoma; Recurrent Malignant Neoplasm; Refractory Classic Hodgkin Lymphoma; Refractory Malignant Neoplasm; Stage III Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Unresectable Melanoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; HIV Infections; Sarcoma, Kaposi; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Melanoma; Lymphoma, Non-Hodgkin; Recurrence; Neoplasms; Lung Neoplasms | interventions — Antiretroviral Therapy, Highly Active; Biopsy; Specimen Handling; pembrolizumab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (pembrolizumab and cART) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Patients continue receiving their recommended combination antiretroviral therapy PO QD. Cycles repeat every 21 days for up to 2 years or 35 doses in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or PET/CT and blood sample collection throughout the trial. Patients may also undergo biopsies during screening and on study.
  Interventions: Drug: Antiretroviral Therapy; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Pembrolizumab; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: Antiretroviral Therapy — Given PO
  Other Names: Anti-Retroviral Therapy; ART
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; QL2107; SCH 900475; SCH-900475; SCH900475
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase I trial studies the side effects of pembrolizumab in treating patients with human immunodeficiency virus (HIV) and malignant neoplasms that have come back (relapsed), do not respond to treatment (refractory), or have distributed over a large area in the body (disseminated). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of MK-3475 (pembrolizumab) in HIV-infected patients on effective antiretroviral therapy and with relapsed/refractory or disseminated acquired immune deficiency syndrome (AIDS)-defining or non-AIDS defining malignancy.

II. To assess the safety and feasibility of MK-3475 (pembrolizumab) administration as first systemic therapy for HIV associated Kaposi sarcoma in patients on effective antiretroviral therapy.

SECONDARY OBJECTIVES:

I. To obtain preliminary insights into clinical benefit (e.g., tumor shrinkage or stabilization >= 24 weeks) across a variety of tumors in patients infected with HIV and on effective antiretroviral therapy.

II. To evaluate the response rate in Kaposi sarcoma impacting physical and/or psychological wellbeing and not amenable to local therapy.

EXPLORATORY OBJECTIVES:

I. To assess the correlation of pre-therapy tumor PD-L1 expression and T-cell infiltration on clinical benefit.

II. To assess the effect of MK-3475 (pembrolizumab) on circulating HIV and the HIV viral reservoir in patients on effective combination anti-retroviral therapy (cART), as measured by plasma HIV single copy ribonucleic acid (RNA), CD4+ T-cell associated HIV unspliced RNA, CD4+ T-cell associated integrated HIV deoxyribonucleic acid (DNA) provirus, ratio of HIV unspliced RNA/DNA, "Tat/Rev induced limiting dilution assay" (TILDA), and phylogenetic analysis of HIV-1 molecular evolution.

III. To evaluate the effect of MK-3475 (pembrolizumab) on host gene expression in circulating blood cells.

IV. To evaluate the effect of MK-3475 (pembrolizumab) on circulating HIV-specific CD8+ T-cell cytotoxicity against autologous HIV infected CD4+ T-cells in patients on effective antiretroviral therapy.

V. To evaluate the effect of MK-3475 (pembrolizumab) on circulating lymphocyte and monocyte numbers and phenotypes.

VI. To assess biopsied tumors from participants that progress by immunohistochemistry arrays and gene expression analysis to evaluate potential reasons for the lack of response to MK-3475 (pembrolizumab) or progression such as a lack of T cells within or around tumor.

VII. To evaluate the effect of pembrolizumab on human herpesvirus 8 (KSHV) viral load in the blood, KSHV seroreactivity and KSHV specific CD8+ T-cell activity.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Patients continue receiving their recommended combination antiretroviral therapy orally (PO) once daily (QD). Cycles repeat every 21 days for up to 2 years or 35 doses in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or positron emission tomography (PET)/CT and blood sample collection throughout the trial. Patients may also undergo biopsies during screening and on study.

After completion of study treatment, patients are followed up 30 days and then every 12 weeks up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven metastatic or locally advanced tumors for which no standard therapy exists, or where standard therapy has failed, or in patients otherwise ineligible for standard therapy, or for an indication that anti-PD-1 therapy has been shown to be effective in studies in HIV-uninfected participants; disease-specific criteria will be applied for certain common cancers and cancers strongly associated with HIV; however, enrollment will not be confined to these tumors
* Non-small cell lung cancer (NSCLC)

  * Metastatic or locally advanced disease that progressed after at least one prior therapy
  * Note: patients that have actionable molecular targets (e.g., epidermal growth factor receptor [EGFR], anaplastic lymphoma kinase [ALK], c-ros oncogene 1[ROS1] mutations) must have received (when indicated) prior appropriate targeted therapy using Food and Drug Administration (FDA)-approved agents
* AIDS-related non-Hodgkin lymphoma and other non-Hodgkin lymphoma

  * Failed standard first-line therapy; and
  * Failed autologous stem cell transplant if indicated for histology (i.e diffuse large B-cell lymphoma) or autologous stem cell transplant is not feasible
* Classical Hodgkin lymphoma

  * Relapsed or refractory de novo classical Hodgkin lymphoma having failed standard first-line therapy; and
  * May have failed to achieve a response or progressed after treatment with brentuximab vedotin or may be brentuximab vedotin naive but is ineligible or unable to receive brentuximab vedotin; and
  * May have failed to achieve a response to, progressed after, or is ineligible for autologous stem cell transplant (auto-SCT)
* Hepatocellular carcinoma (HCC)

  * Not eligible for curative attempt resection or liver transplant
* Kaposi sarcoma impacting physical and/or psychological wellbeing and not amenable to local therapy. Patients who have received prior therapy and treatment naive patients are both potentially eligible to participate.

  * On antiretrovival therapy (ART) with suppressed HIV viral load for > 3 months (Note: an extended washout period is needed to avoid treatment during the period of risk for the highly toxic and often fatal "Immune Reconstitution Inflammatory Syndrome (IRIS)"
  * No KSHV-associated multicentric Castleman disease in past 5 years
  * No symptomatic pulmonary Kapsoi sarcoma (KS) or chest X-rays positive for un-evaluated abnormalities
  * Disease evaluable by AIDS Clinical Trial Group (ACTG) KS response criteria
  * CD4+ T-cell count >= 50 cells/uL
  * For KS patients, the following laboratory values supersede values below:

    * Platelets > lower limit of normal
    * Hemoglobin > 10 g/dL
* Melanoma

  * Unresectable or metastatic disease progression following a BRAF inhibitor if BRAF V600 positive
  * Note: Prior therapy with ipilimumab not required
* Available pretreatment biopsy, either fresh (optimal) or archival (acceptable)
* Resolution of any adverse events (AEs) from prior treatments must be resolved to baseline or grade =< 1 at enrollment (with the exception of alopecia), neuropathy, and ototoxicity (i.e., AEs that are not expected to improve within the washout period)
* On an effective combination cART regimen, generally a 3-drug regimen based on Department of Health and Human Services (DHHS) treatment guidelines

  * Patients must be on cART >= 4 weeks; and
  * Evidence of viral suppression defined as HIV viral load < 200 copies/mL; and
  * No symptomatic AEs > grade 1 by Common Terminology Criteria for Adverse Events (CTCAE) criteria probably or definitely attributed to cART; and
  * No laboratory AEs noted on protocol defined screening laboratories > grade 1 by CTCAE criteria probably or definitely attributed to cART, with exceptions noted below
  * Note: if cART is modified during the screening period, patients must be on an effective new regimen for >= 2 weeks and otherwise meet eligibility criteria
  * Most patients have viral loads that are suppressible to < 50 copies/mL, but about 25% of patients will occasionally have blips up to 400-500 copies/mL, which do not appear to correlate with lack of viral suppression in most studies; thus, an HIV viral load of =< 400 copies/mL for an occasional "blip" will be allowed, if there is documentation of an HIV viral load < 200 on the same regimen and no significant treatment interruption
* CD4+ T-cell count >= 50 cells/uL
* Patients must have marrow function and organ function as defined below

  * Note: to remain on treatment, any abnormal lab values allowed by the PI must remain stable or improve during treatment; similar off treatment rules will be applied to all patients, except the following: the grade of any abnormal laboratory (lab) value allowed by the protocol principal investigator (PI) at enrollment will be considered the patient's baseline for potentially resuming therapy after modification/holding of therapy when off treatment criteria are applied
* Leukocytes no lower limit
* Absolute neutrophil count > 500/mcL
* Platelets > 50,000/mcL
* Hemoglobin > 9 g/dL
* Total bilirubin < 1.5 X upper limit of normal (ULN); or < 3 x institutional ULN for Gilbert's syndrome or HIV protease inhibitors; or < 5 x ULN and direct bilirubin < 0.7 mg/dL for patients on atazanavir containing HIV regimen
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 X institutional ULN
* Creatine kinase < 5 X institutional ULN
* Serum creatinine < 2.5 X institutional ULN OR measured or calculated* creatinine clearance (CrCl) (glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl) >= 30 mL/min for subject with creatinine levels > 2.5 X institutional ULN

  * Creatinine clearance should be calculated per institutional standard
* Thyroid stimulating hormone (TSH) within institutional limits (ie: normal); if TSH is greater or less than institutional limits patients may participate if their T4 is within normal limits (WNL); patients may be on a stable dose of replacement thyroid medication; dose adjustments are allowed if needed
* Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 1
* At least 2 weeks from end of chemotherapy with resolution of neutropenia to above level
* At least 2 weeks from end of radiation therapy
* At least 4 weeks from end of monoclonal antibody therapy
* At least 2 weeks from end of targeted therapy
* Female patients of childbearing potential must have a negative urine or serum pregnancy within 72 hours before receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required

  * Note: the effects of MK-3475 on the developing human fetus are unknown; for this reason and because anti-PD-1 agents may be teratogenic, women of child-bearing potential must agree to use 2 methods of birth control, or be surgically sterile, or abstain from heterosexual activity beginning with the screening visit and for the duration of study participation, through 120 days beyond last dose of MK-3475 administration; patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
  * Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Men treated or enrolled on this protocol must agree to use 2 adequate methods of contraception starting with the screening visit, for the duration of study participation, and through 120 days after the last dose of MK-3475 administration
* No prior treatment with anti-PD-1 or anti-PD-L1
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 or other tumor-specific criteria or disease assessable by physical exam or other methods if not measurable by RECIST
* Baseline tumor tissue, either fresh (preferred) or from paraffin block/unstained slides if contemporary biopsy is unsafe or not otherwise obtainable from the primary tumor site or metastatic site to be available for use on correlative studies
* Age >= 18 years

  * Because no dosing or adverse event data are currently available on the use of MK-3475 (pembrolizumab) in combination with cART in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Active systemic immunosuppressive therapy
* Systemic steroid therapy or steroid therapy that cannot be discontinued with more than 7 consecutive days of steroids within the prior 2 weeks

  * Note: the use of prednisone or equivalent < 0.125 mg/kg/day (absolute maximum of 15 mg/day) as replacement therapy is permitted; inhaled or topical corticosteroids are permitted
* Current or history of systemic autoimmune disease requiring systemic therapy

  * Note: the following will NOT be exclusionary:

    * The presence of laboratory evidence of autoimmune disease (e.g., positive antinuclear antibody [ANA] titer or lupus anticoagulant) without associated symptoms
    * Clinical evidence of vitiligo or other forms of depigmenting illness
    * Mild autoimmunity not impacting the function of major organs (e.g., limited psoriasis)
* Grade 3 or 4 immune related toxicity associated with prior ipilimumab therapy that has not resolved to grade 0 or 1
* Cardiovascular disease that meets one of the following: congestive heart failure (New York Heart Association class III or IV), active angina pectoris, or recent myocardial infarction (within the last 6 months)
* Active tuberculosis (TB) or atypical mycobacterial infection:

  * Patients who are undergoing systemic antibiotics for active mycobacterial infection
  * Patients with TB immune reconstitution syndrome (IRIS) requiring corticosteroids

    * Note: patients who are receiving treatment for latent tuberculosis (isonicotinylhydrazide [INH] or alternative) may be eligible after discussion with the protocol P.I.
* Cirrhosis with Child-Pugh score of B or C
* Uncontrolled hepatitis B virus (HBV) infection, defined as acute liver failure or protracted, severe course, as indicated by total bilirubin > 3 mg/dL (or direct bilirubin > 1.5 mg/dL), international normalized ratio > 1.5, encephalopathy, or ascites

  * Note: the following will NOT be exclusionary:

    * A positive hepatitis B serology indicative of previous immunization (i.e., hepatitis B surface antibody [HBsAb] positive and hepatitis B core antibody [HBcAb] negative), or a fully resolved acute HBV infection
    * Patients with chronic HBV infection suppressed by appropriate antiretroviral therapy with activity against HBV, as outlined in DHHS guidelines
* Uncontrolled hepatitis C virus (HCV) infection, defined as plasma HCV RNA detectable by PCR

  * Note: the following will NOT be exclusionary:

    * Positive HCV serology but no detectable HCV RNA, indicative of spontaneously cleared HCV infection
    * Patients who have been successfully treated for HCV as long as therapy for HCV has been completed
* Patients who are receiving any other investigational agents for cancer
* Extensive active brain disease including symptomatic brain metastases or the presence of leptomeningeal disease, and all patients with infratentorial tumors

  * Note: patients with brain metastasis after definitive therapy with surgery or stereotactic radiation and stable off steroids for > 4 weeks are eligible as are patients with asymptomatic brain metastasis as long as less than 1 cm and thus deemed as not requiring therapy by the primary physician and the lesions(s) are not infratentorial
* Pregnancy or nursing or unwilling to take adequate birth control during therapy
* Prior organ allograft or allogeneic transplantation, if the transplanted tissue is still in place
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia
* Medical or psychiatric illness or social situations that would, in the opinion of the investigator, preclude participation in the study or the ability of patients to provide informed consent for themselves
* Clinically significant lung disease including known history or evidence of interstitial lung disease or chronic obstructive pulmonary disease (COPD) that requires oxygen therapy
* Active non-infectious pneumonitis >= grade 2 or history of grade 3 non-infectious pneumonitis requiring steroids within the past 12 months; or any history of grade 4 non-infectious pneumonitis
* Grade 3-4 ascites or pleural effusion

  * Note: The following will NOT be exclusionary: A participant who is clinically stable following treatment for ascites or pleural effusion (including therapeutic thoracentesis or paracentesis)
* Receipt of live vaccines within 30 days before the first dose of trial treatment and while participating in the trial; examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, seasonal flu, H1N1 flu, rabies, bacillus Calmette-Guerin (BCG), and typhoid vaccine
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-3475 (pembrolizumab)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2024-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Lurain, Principal Investigator — Cancer Immunotherapy Trials Network
Locations (12):
- United States (12):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - FHCC South Lake Union, Seattle, Washington

REFERENCES:
- [Derived] Lurain K, Ramaswami R, Ekwede I, Eulo V, Goyal G, Menon M, Odeny TA, Sharon E, Wagner MJ, Wang CJ, Bhardwaj N, Friedlander PA, Abdul-Hay M, Cornejo Castro EM, Labo N, Marshall VA, Miley W, Moore K, Roshan R, Whitby D, Kask AS, Kaiser J, Han E, Wright A, Yarchoan R, Fling SP, Uldrick TS. Cancer Immunotherapy Trials Network 12: Pembrolizumab in HIV-Associated Kaposi Sarcoma. J Clin Oncol. 2025 Feb;43(4):432-442. doi: 10.1200/JCO.24.00640. Epub 2024 Oct 2. PMID 39356983
- [Derived] Uldrick TS, Adams SV, Fromentin R, Roche M, Fling SP, Goncalves PH, Lurain K, Ramaswami R, Wang CJ, Gorelick RJ, Welker JL, O'Donoghue L, Choudhary H, Lifson JD, Rasmussen TA, Rhodes A, Tumpach C, Yarchoan R, Maldarelli F, Cheever MA, Sekaly R, Chomont N, Deeks SG, Lewin SR. Pembrolizumab induces HIV latency reversal in people living with HIV and cancer on antiretroviral therapy. Sci Transl Med. 2022 Jan 26;14(629):eabl3836. doi: 10.1126/scitranslmed.abl3836. Epub 2022 Jan 26. PMID 35080914
- [Derived] Uldrick TS, Goncalves PH, Abdul-Hay M, Claeys AJ, Emu B, Ernstoff MS, Fling SP, Fong L, Kaiser JC, Lacroix AM, Lee SY, Lundgren LM, Lurain K, Parsons CH, Peeramsetti S, Ramaswami R, Sharon E, Sznol M, Wang CJ, Yarchoan R, Cheever MA; Cancer Immunotherapy Trials Network (CITN)-12 Study Team. Assessment of the Safety of Pembrolizumab in Patients With HIV and Advanced Cancer-A Phase 1 Study. JAMA Oncol. 2019 Sep 1;5(9):1332-1339. doi: 10.1001/jamaoncol.2019.2244. PMID 31154457

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per the protocol, participants enrolled into Cohorts 1-3 were combined into one group for analysis. The number of participants enrolled to each cohort was not sufficient to perform subgroup analysis based on a CD4 count.
Groups:
- Cohorts 1-3 (Pembrolizumab and cART): Participants enrolled into 1 of 3 cohorts based on CD4+ T-cell counts, who receive pembrolizumab IV over 30 minutes on day 1. Participants continue receiving their recommended combination antiretroviral therapy (cART) per established regimen. Cycles repeat every 21 days for up to 2 years or 35 doses in the absence of disease progression or unacceptable toxicity. Participants also undergo CT or PET/CT and blood sample collection throughout the trial. Participants may also undergo biopsies during screening and on study.
  Antiretroviral Therapy: Given PO
  Biopsy: Undergo biopsy
  Biospecimen Collection: Undergo blood sample collection
  Computed Tomography: Undergo CT or PET/CT
  Pembrolizumab: Given IV
  Positron Emission Tomography: Undergo PET/CT
- Cohort 4 (Pembrolizumab and cART): Participants with HIV associated Kaposi Sarcoma enrolled into cohort 4, who receive pembrolizumab IV over 30 minutes on day 1. Participants continue receiving their recommended combination antiretroviral therapy (cART) per established regimen. Cycles repeat every 21 days for up to 2 years or 35 doses in the absence of disease progression or unacceptable toxicity. Participants also undergo CT or PET/CT and blood sample collection throughout the trial. Participants may also undergo biopsies during screening and on study.
  Antiretroviral Therapy: Given PO
  Biopsy: Undergo biopsy
  Biospecimen Collection: Undergo blood sample collection
  Computed Tomography: Undergo CT or PET/CT
  Pembrolizumab: Given IV
  Positron Emission Tomography: Undergo PET/CT
Period: Overall Study
Arm/Group | Cohorts 1-3 (Pembrolizumab and cART) | Cohort 4 (Pembrolizumab and cART)
Started | 34 | 24
Completed (Participants who completed 2 years or 35 cycles of study treatment.) | 2 | 2
Not Completed | 32 | 22
Not completed — Adverse Event | 2 | 5
Not completed — Complicating Disease/Intercurrent Illness | 1 | 1
Not completed — Death | 0 | 1
Not completed — Incarceration | 1 | 0
Not completed — Lack of Efficacy | 17 | 7
Not completed — Physician Decision | 4 | 3
Not completed — Switched to Alternative Treatment | 1 | 0
Not completed — Study Terminated | 0 | 4
Not completed — Withdrawal by Subject | 6 | 1

BASELINE CHARACTERISTICS:
Population: Participants do not have to complete the study in order to be included in the analysis population for the primary outcome measure.
Groups:
- Cohorts 1-3 (Pembrolizumab and cART): Participants enrolled into 1 of 3 cohorts based on CD4+ T-cell counts, who receive pembrolizumab IV over 30 minutes on day 1. Participants continue receiving their recommended combination antiretroviral therapy per established regimen. Cycles repeat every 21 days for up to 2 years or 35 doses in the absence of disease progression or unacceptable toxicity. Participants also undergo CT or PET/CT and blood sample collection throughout the trial. Participants may also undergo biopsies during screening and on study.
  Per the protocol, participants enrolled into Cohorts 1-3 were combined into one group for analysis. The number of participants enrolled to each cohort (n=12) was not sufficient to perform subgroup analysis based on a CD4 count
  Antiretroviral Therapy: Given PO
  Biopsy: Undergo biopsy
  Biospecimen Collection: Undergo blood sample collection
  Computed Tomography: Undergo CT or PET/CT
  Pembrolizumab: Given IV
  Positron Emission Tomography: Undergo PET/CT
- Cohort 4 (Pembrolizumab and cART): Participants with HIV associated Kaposi sarcoma enrolled into cohort 4, who receive pembrolizumab IV over 30 minutes on day 1. Participants continue receiving their recommended combination antiretroviral therapy per established regimen. Cycles repeat every 21 days for up to 2 years or 35 doses in the absence of disease progression or unacceptable toxicity. Participants also undergo CT or PET/CT and blood sample collection throughout the trial. Participants may also undergo biopsies during screening and on study.
  Antiretroviral Therapy: Given PO
  Biopsy: Undergo biopsy
  Biospecimen Collection: Undergo blood sample collection
  Computed Tomography: Undergo CT or PET/CT
  Pembrolizumab: Given IV
  Positron Emission Tomography: Undergo PET/CT
- Total: Total of all reporting groups
Arm/Group | Cohorts 1-3 (Pembrolizumab and cART) | Cohort 4 (Pembrolizumab and cART) | Total
Number analyzed (Participants) | 34 | 24 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 23 | 51
  >=65 years | 6 | 1 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (9.3) | 44.5 (10.7) | 51.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 30 | 24 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 30 | 19 | 49
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 10 | 13 | 23
  White | 20 | 10 | 30
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 34 | 24 | 58
MK-3475 (Pembrolizumab) as First Systemic Therapy [Count of Participants; unit: Participants] | 26 | 9 | 35

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Observed Adverse Events (AEs)
Description: Will be graded using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (version 5.0 beginning April 1, 2018). Safety and tolerability will be assessed by summarizing all relevant parameters including AEs, serious AEs, laboratory tests, vital signs, and electrocardiogram measurements. All summaries will be presented for each cohort and overall. If the numbers are sufficient, the results may additionally be stratified by tumor type.
Time Frame: Up to 90 days after the last dose of trial treatment, up to 2 years or 35 cycles of trial treatment.
Population: Participants who received at least 1 dose of the study drug.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 1 (Pembrolizumab and cART): Participants enrolled into Cohort 1 (50-199 CD4+ T cells/mcL), who receive pembrolizumab IV over 30 minutes on day 1. Participants continue receiving their recommended combination antiretroviral therapy per established regimen. Cycles repeat every 21 days for up to 2 years or 35 doses in the absence of disease progression or unacceptable toxicity. Participants also undergo CT or PET/CT and blood sample collection throughout the trial. Participants may also undergo biopsies during screening and on study.
  Antiretroviral Therapy: Given PO
  Biopsy: Undergo biopsy
  Biospecimen Collection: Undergo blood sample collection
  Computed Tomography: Undergo CT or PET/CT
  Pembrolizumab: Given IV
  Positron Emission Tomography: Undergo PET/CT
- Cohort 2 (Pembrolizumab and cART): Participants enrolled into Cohort 2 (200-350 CD4+ cells/mcL), who receive pembrolizumab IV over 30 minutes on day 1. Participants continue receiving their recommended combination antiretroviral therapy per established regimen. Cycles repeat every 21 days for up to 2 years or 35 doses in the absence of disease progression or unacceptable toxicity. Participants also undergo CT or PET/CT and blood sample collection throughout the trial. Participants may also undergo biopsies during screening and on study.
  Antiretroviral Therapy: Given PO
  Biopsy: Undergo biopsy
  Biospecimen Collection: Undergo blood sample collection
  Computed Tomography: Undergo CT or PET/CT
  Pembrolizumab: Given IV
  Positron Emission Tomography: Undergo PET/CT
- Cohort 3 (Pembrolizumab and cART): Participants enrolled into Cohort 3 (> 350 CD4+ cells/mcl), who receive pembrolizumab IV over 30 minutes on day 1. Participants continue receiving their recommended combination antiretroviral therapy per established regimen. Cycles repeat every 21 days for up to 2 years or 35 doses in the absence of disease progression or unacceptable toxicity. Participants also undergo CT or PET/CT and blood sample collection throughout the trial. Participants may also undergo biopsies during screening and on study.
  Antiretroviral Therapy: Given PO
  Biopsy: Undergo biopsy
  Biospecimen Collection: Undergo blood sample collection
  Computed Tomography: Undergo CT or PET/CT
  Pembrolizumab: Given IV
  Positron Emission Tomography: Undergo PET/CT
- Cohort 4 (Pembrolizumab and cART): Participants with HIV associated Kaposi sarcoma enrolled into cohort 4, who receive pembrolizumab IV over 30 minutes on day 1. Participants continue receiving their recommended combination antiretroviral therapy per established regimen. Cycles repeat every 21 days for up to 2 years or 35 doses in the absence of disease progression or unacceptable toxicity. Participants undergo physical examination and blood sample collection, and may undergo CT or PET/CT. Participants may also undergo biopsies during screening and on study.
  Antiretroviral Therapy: Given PO
  Biopsy: Undergo biopsy
  Biospecimen Collection: Undergo blood sample collection
  Computed Tomography: Undergo CT or PET/CT
  Pembrolizumab: Given IV
  Positron Emission Tomography: Undergo PET/CT
- Total: Participants enrolled into Cohorts 1-4, who receive pembrolizumab IV over 30 minutes on day 1. Participants continue receiving their recommended combination antiretroviral therapy per established regimen. Cycles repeat every 21 days for up to 2 years or 35 doses in the absence of disease progression or unacceptable toxicity. Participants also undergo physical examination, CT or PET/CT, and blood sample collection throughout the trial. Participants may also undergo biopsies during screening and on study.
  Antiretroviral Therapy: Given PO
  Biopsy: Undergo biopsy
  Biospecimen Collection: Undergo blood sample collection
  Computed Tomography: Undergo CT or PET/CT
  Pembrolizumab: Given IV
  Positron Emission Tomography: Undergo PET/CT
Arm/Group | Cohort 1 (Pembrolizumab and cART) | Cohort 2 (Pembrolizumab and cART) | Cohort 3 (Pembrolizumab and cART) | Cohort 4 (Pembrolizumab and cART) | Total
Number analyzed (Participants) | 10 | 12 | 12 | 24 | 58
percentage of participants | 100 | 100 | 100 | 100 | 100

2. Primary Outcome: Incidence of Immune-related Events of Clinical Interest (irECI)
Description: This includes the occurrence of grade 2 or higher AEs. Will be graded using CTCAE version 4.0 (version 5.0 beginning April 1, 2018). Any AE of unknown etiology associated with study therapy will be evaluated to determine if it is possibly an ECI of a potentially immunologic etiology or related to combination antiretroviral therapy (cART). All summaries will be presented for each cohort and overall. If the numbers are sufficient, the results may additionally be stratified by tumor type.
Time Frame: Up to 90 days after the last dose of trial treatment, up to 2 years or 35 cycles of trial treatment.
Population: Participants who received at least 1 dose of the study drug
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (Pembrolizumab and cART) | Cohort 2 (Pembrolizumab and cART) | Cohort 3 (Pembrolizumab and cART) | Cohort 4 (Pembrolizumab and cART) | Total
Number analyzed (Participants) | 10 | 12 | 12 | 24 | 58
percentage of participants | 20.0 | 50.0 | 25.0 | 20.8 | 27.6

3. Primary Outcome: Incidence of cART-related ECIs of Grade 2 or Higher AEs
Description: Will be graded using CTCAE version 4.0 (version 5.0 beginning April 1, 2018). Any AE of unknown etiology associated with study therapy will be evaluated to determine if it is possibly an ECI of a potentially immunologic etiology or related to cART. All summaries will be presented for each cohort and overall. If the numbers are sufficient, the results may additionally be stratified by tumor type.
Time Frame: Up to 90 days after the last dose of trial treatment, up to 2 years or 35 cycles of trial treatment.
Population: Participants who received at least 1 dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (Pembrolizumab and cART) | Cohort 2 (Pembrolizumab and cART) | Cohort 3 (Pembrolizumab and cART) | Cohort 4 (Pembrolizumab and cART) | Total
Number analyzed (Participants) | 10 | 12 | 12 | 24 | 58
percentage of participants | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Objective Response Rate (Cohorts 1-3)
Description: Defined as the proportion of participants who achieved complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, "Lugano Criteria" for Malignant Lymphoma or other tumor-specific criteria. Analyzed using Clopper-Pearson 95% confidence intervals.
Time Frame: Up to 2 years
Population: Analysis is based on all participants who have received at least one dose of study treatment. Participants with missing outcomes considered nonresponders. Participants without progression were censored at the last disease assessment date.
  Per the protocol, participants enrolled into Cohorts 1-3 were combined into one group for analysis. The number of participants enrolled to each cohort was not sufficient to perform subgroup analysis based on a CD4 count.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohorts 1-3 (Pembrolizumab and cART): Participants enrolled into 1 of 3 cohorts based on CD4+ T-cell counts, who receive pembrolizumab IV over 30 minutes on day 1. Participants continue receiving their recommended combination antiretroviral therapy per established regimen. Cycles repeat every 21 days for up to 2 years or 35 doses in the absence of disease progression or unacceptable toxicity. Participants also undergo CT or PET/CT and blood sample collection throughout the trial. Participants may also undergo biopsies during screening and on study.
  Antiretroviral Therapy: Given PO
  Biopsy: Undergo biopsy
  Biospecimen Collection: Undergo blood sample collection
  Computed Tomography: Undergo CT or PET/CT
  Pembrolizumab: Given IV
  Positron Emission Tomography: Undergo PET/CT
Arm/Group | Cohorts 1-3 (Pembrolizumab and cART)
Number analyzed (Participants) | 34
percentage of participants | 14.7 [5.0 to 31.1]

5. Secondary Outcome: Progression-free Survival (Cohorts 1-3)
Description: Assessed using RECIST 1.1, "Lugano Criteria" for Malignant Lymphoma or other tumor-specific criteria. Summarized statistically using Kaplan-Meier method.
Time Frame: From the first dose of study drug to progressive disease or death, whichever occurs earlier, assessed up to 25 months
Population: All participants who receive at least one dose of study drug. Participants without documented progressive disease or death will be censored at the last disease assessment date.
  Per the protocol, participants enrolled into Cohorts 1-3 were combined into one group for analysis. The number of participants enrolled to each cohort was not sufficient to perform subgroup analysis based on a CD4 count.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohorts 1-3 (Pembrolizumab and cART)
Number analyzed (Participants) | 34
months | 3.9 [2.8 to 4.8]

6. Secondary Outcome: Duration of Response (Cohorts 1-3)
Description: Defined in participants experiencing CR or PR using RECIST 1.1, "Lugano Criteria" for malignant lymphoma or other tumor-specific criteria. Summarized statistically using Kaplan-Meier method.
Time Frame: Interval between the date of first response (CR/PR) and the date of progression, assessed up to 2 years
Population: Analysis is based on all participants who received at least one dose of study drug. Participants without documented progression were censored at the last disease assessment date.
  Per the protocol, participants enrolled into Cohorts 1-3 were combined into one group for analysis. The number of participants enrolled to each cohort was not sufficient to perform subgroup analysis based on a CD4 count.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Cohorts 1-3 (Pembrolizumab and cART): Patients enrolled into 1 of 3 cohorts based on CD4+ T-cell counts, who receive pembrolizumab IV over 30 minutes on day 1. Patients continue receiving their recommended combination antiretroviral therapy per established regimen. Cycles repeat every 21 days for up to 2 years or 35 doses in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or PET/CT and blood sample collection throughout the trial. Patients may also undergo biopsies during screening and on study.
  Antiretroviral Therapy: Given PO
  Biopsy: Undergo biopsy
  Biospecimen Collection: Undergo blood sample collection
  Computed Tomography: Undergo CT or PET/CT
  Pembrolizumab: Given IV
  Positron Emission Tomography: Undergo PET/CT
Arm/Group | Cohorts 1-3 (Pembrolizumab and cART)
Number analyzed (Participants) | 34
months | NA [NA to NA] — Median duration of response (DOR) could not be calculated. Upper and lower confidence interval for DOR could not be obtained using Kaplan-Meier estimates. Insufficient number of participants with events.

7. Secondary Outcome: Overall Survival (Cohorts 1-3)
Description: Summarized statistically using Kaplan-Meier method.
Time Frame: From the first dose of study drug to death due to any cause, assessed up to 3 years
Population: Participants who receive at least one dose of study drug. Participants without documented death at the time of analysis were censored at the date last known to be alive.
  Per the protocol, participants enrolled into Cohorts 1-3 were combined into one group for analysis. The number of participants enrolled to each cohort was not sufficient to perform subgroup analysis based on a CD4 count.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohorts 1-3 (Pembrolizumab and cART)
Number analyzed (Participants) | 34
months | 14.5 [11.5 to 21.3]

8. Secondary Outcome: Objective Response Rate (Partial Response + Completion Response)(Kaposi Sarcoma Cohort)
Description: Defined as the proportion of participants who achieved the best objective response rate (complete response (CR) + partial response (PR)) as determined by modified Acquired Immunodeficiency Syndrome Clinical Trials Group (ACTG) criteria Analyzed using Clopper-Pearson 95% confidence intervals.
Time Frame: Up to 2 years
Population: Analysis is based on all participants who have received at least one dose of study treatment. Participants with missing outcomes considered nonresponders. Participants without progression were censored at the last disease assessment date.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Kaposi Sarcoma Cohort (Pembrolizumab and cART): Participants enrolled into Cohort 4 and participants with evaluable HIV associated Kaposi sarcoma enrolled into Cohorts 1-3, who receive pembrolizumab IV over 30 minutes on day 1. Participants continue receiving their recommended combination antiretroviral therapy per established regimen. Cycles repeat every 21 days for up to 2 years or 35 doses in the absence of disease progression or unacceptable toxicity. Participants undergo physical examination and blood sample collection, and may undergo CT or PET/CT. Participants may also undergo biopsies during screening and on study.
  Antiretroviral Therapy: Given PO
  Biopsy: Undergo biopsy
  Biospecimen Collection: Undergo blood sample collection
  Computed Tomography: Undergo CT or PET/CT
  Pembrolizumab: Given IV
  Positron Emission Tomography: Undergo PET/CT
- Treatment Naïve Kaposi Sarcoma Cohort (Pembrolizumab and cART): Treatment naïve participants enrolled into Cohort 4 and treatment naïve participants with evaluable HIV associated Kaposi sarcoma enrolled into Cohorts 1-3, who receive pembrolizumab IV over 30 minutes on day 1. Participants continue receiving their recommended combination antiretroviral therapy per established regimen. Cycles repeat every 21 days for up to 2 years or 35 doses in the absence of disease progression or unacceptable toxicity. Participants undergo physical examination and blood sample collection, and may undergo CT or PET/CT. Participants may also undergo biopsies during screening and on study.
  Antiretroviral Therapy: Given PO
  Biopsy: Undergo biopsy
  Biospecimen Collection: Undergo blood sample collection
  Computed Tomography: Undergo CT or PET/CT
  Pembrolizumab: Given IV
  Positron Emission Tomography: Undergo PET/CT
- Previously Treated Kaposi Sarcoma Cohort (Pembrolizumab and cART): Previously treated participants enrolled into Cohort 4 and previously treated participants with evaluable HIV associated Kaposi sarcoma enrolled into Cohorts 1-3, who receive pembrolizumab IV over 30 minutes on day 1. Participants continue receiving their recommended combination antiretroviral therapy per established regimen. Cycles repeat every 21 days for up to 2 years or 35 doses in the absence of disease progression or unacceptable toxicity. Participants undergo physical examination and blood sample collection, and may undergo CT or PET/CT. Participants may also undergo biopsies during screening and on study.
  Antiretroviral Therapy: Given PO
  Biopsy: Undergo biopsy
  Biospecimen Collection: Undergo blood sample collection
  Computed Tomography: Undergo CT or PET/CT
  Pembrolizumab: Given IV
  Positron Emission Tomography: Undergo PET/CT
Arm/Group | Kaposi Sarcoma Cohort (Pembrolizumab and cART) | Treatment Naïve Kaposi Sarcoma Cohort (Pembrolizumab and cART) | Previously Treated Kaposi Sarcoma Cohort (Pembrolizumab and cART)
Number analyzed (Participants) | 29 | 8 | 21
percentage of participants | 62.1 [42.3 to 79.3] | 87.5 [47.3 to 99.7] | 52.4 [29.8 to 74.3]

9. Secondary Outcome: Progression-free Survival (Kaposi Sarcoma Cohort)
Description: Assessed using ACTG criteria. Summarized statistically using Kaplan-Meier method.
Time Frame: From the first dose of study drug to progressive disease or death, whichever occurs earlier, assessed up to 3 years
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Kaposi Sarcoma Cohort (Pembrolizumab and cART) | Treatment Naïve Kaposi Sarcoma Cohort (Pembrolizumab and cART) | Previously Treated Kaposi Sarcoma Cohort (Pembrolizumab and cART)
Number analyzed (Participants) | 29 | 8 | 21
months | 28.2 [4.2 to NA] — Upper confidence interval for PFS could not be obtained based on Kaplan-Meier estimates. Insufficient number of participants with events. | 28.2 [3.3 to NA] — Upper confidence interval for PFS could not be obtained based on Kaplan-Meier estimates. Insufficient number of participants with events. | NA [2.8 to NA] — Median PFS could not be calculated and upper confidence interval was not obtained based on Kaplan-Meier estimates. Insufficient number of participants with events.

10. Secondary Outcome: Duration of Response (Kaposi Sarcoma Cohort)
Description: Assessed using ACTG criteria. Summarized statistically using Kaplan-Meier method.
Time Frame: Interval between the date of first response (CR/PR) and the date of progression, assessed up to 2 years
Population: Analysis is based on all participants who received at least one dose of study drug. Participants without documented progression were censored at the last disease assessment date.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Kaposi Sarcoma Cohort (Pembrolizumab and cART) | Treatment Naïve Kaposi Sarcoma Cohort (Pembrolizumab and cART) | Previously Treated Kaposi Sarcoma Cohort (Pembrolizumab and cART)
Number analyzed (Participants) | 29 | 8 | 21
months | NA [NA to NA] — Median for duration of response (DOR) was not calculated. Lower and upper confidence intervals for DOR were not obtained based on the Kaplan-Meier estimates. Insufficient number of participants with events. | NA [3.5 to NA] — Median for duration of response (DOR) was not calculated. Upper confidence interval for DOR were not obtained based on the Kaplan-Meier estimates. Insufficient number of participants with events. | NA [NA to NA] — Median for duration of response was not calculated. Lower and upper confidence intervals for DOR were not obtained based on the Kaplan-Meier estimates. Insufficient number of participants with events.

11. Secondary Outcome: Overall Survival (Kaposi Sarcoma Cohort)
Description: Summarized statistically using Kaplan-Meier method.
Time Frame: From the first dose of study drug to death due to any cause, assessed up to 3 years
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Kaposi Sarcoma Cohort (Pembrolizumab and cART): Participants enrolled into Cohort 4 and participants with HIV associated Kaposi sarcoma enrolled into Cohorts 1-3, who receive pembrolizumab IV over 30 minutes on day 1. Participants continue receiving their recommended combination antiretroviral therapy per established regimen. Cycles repeat every 21 days for up to 2 years or 35 doses in the absence of disease progression or unacceptable toxicity. Participants undergo physical examination and blood sample collection, and may undergo CT or PET/CT. Participants may also undergo biopsies during screening and on study.
  Antiretroviral Therapy: Given PO
  Biopsy: Undergo biopsy
  Biospecimen Collection: Undergo blood sample collection
  Computed Tomography: Undergo CT or PET/CT
  Pembrolizumab: Given IV
  Positron Emission Tomography: Undergo PET/CT
- Treatment Naïve Kaposi Sarcoma Cohort (Pembrolizumab and cART): Treatment naïve participants enrolled into Cohort 4 and treatment naïve participants with HIV associated Kaposi sarcoma enrolled into Cohorts 1-3, who receive pembrolizumab IV over 30 minutes on day 1. Participants continue receiving their recommended combination antiretroviral therapy per established regimen. Cycles repeat every 21 days for up to 2 years or 35 doses in the absence of disease progression or unacceptable toxicity. Participants undergo physical examination and blood sample collection, and may undergo CT or PET/CT. Participants may also undergo biopsies during screening and on study.
  Antiretroviral Therapy: Given PO
  Biopsy: Undergo biopsy
  Biospecimen Collection: Undergo blood sample collection
  Computed Tomography: Undergo CT or PET/CT
  Pembrolizumab: Given IV
  Positron Emission Tomography: Undergo PET/CT
Arm/Group | Kaposi Sarcoma Cohort (Pembrolizumab and cART) | Treatment Naïve Kaposi Sarcoma Cohort (Pembrolizumab and cART) | Previously Treated Kaposi Sarcoma Cohort (Pembrolizumab and cART)
Number analyzed (Participants) | 32 | 9 | 23
months | NA [28.2 to NA] — Median survival time could not be calculated and upper limit for the confidence interval were not obtained based on the Kaplan-Meier estimates. Insufficient number of participants with events. | NA [28.2 to NA] — Median survival time could not be calculated and upper limit for the confidence interval were not obtained based on the Kaplan-Meier estimates. Insufficient number of participants with events. | NA [17.2 to NA] — Median survival time could not be calculated and upper limit for the confidence interval were not obtained based on the Kaplan-Meier estimates. Insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: Up to 90 days after the last dose of trial treatment, up to 2 years or 35 cycles of trial treatment. All cause mortality was assessed for up to 36 months.
Description: Will be graded using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (version 5.0 beginning April 1, 2018). Safety and tolerability will be assessed by summarizing all relevant parameters including AEs, serious AEs, laboratory tests, vital signs, and electrocardiogram measurements. All summaries will be presented for each cohort and overall.
Arm/Group | Cohort 1 (Pembrolizumab and cART) | Cohort 2 (Pembrolizumab and cART) | Cohort 3 (Pembrolizumab and cART) | Cohort 4 (Pembrolizumab and cART) | Total
All-Cause Mortality (participants affected / at risk) | 5/10 | 5/12 | 5/12 | 2/24 | 17/58
Serious Adverse Events (participants affected / at risk) | 8/10 | 8/12 | 6/12 | 9/24 | 31/58
Other Adverse Events (participants affected / at risk) | 10/10 | 12/12 | 12/12 | 24/24 | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Pembrolizumab and cART) (N=10) | Cohort 2 (Pembrolizumab and cART) (N=12) | Cohort 3 (Pembrolizumab and cART) (N=12) | Cohort 4 (Pembrolizumab and cART) (N=24) | Total (N=58)
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1 | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Hemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 3 | 6
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Bronchopulmonary hemorrhage - hemoptisis (General disorders) | 1 | 0 | 0 | 0 | 1
Death NOS (General disorders) | 0 | 2 | 0 | 0 | 2
Edema limbs (General disorders) | 0 | 1 | 0 | 0 | 1
Edema trunk (General disorders) | 0 | 1 | 0 | 0 | 1
Failure to thrive (General disorders) | 0 | 1 | 0 | 0 | 1
Fever (General disorders) | 1 | 1 | 1 | 1 | 4
Localized edema (General disorders) | 0 | 1 | 0 | 0 | 1
Non-cardiac chest pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0 | 1
Pulmonary embolism - thromboembolic event (General disorders) | 1 | 0 | 0 | 0 | 1
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Mycobacterium avium complex (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Skin infection (Infections and infestations) | 2 | 0 | 0 | 0 | 2
Soft tissue infection (Infections and infestations) | 0 | 0 | 2 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Creatinine increased (Investigations) | 2 | 1 | 0 | 0 | 3
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 5 | 0 | 0 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Death due to progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Metastatic anal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Prostate cancer progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 2
Other, Disposition Issue (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 3
Proteinurea (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1 | 2
Thromboembolic event (Vascular disorders) | 1 | 0 | 1 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Pembrolizumab and cART) (N=10) | Cohort 2 (Pembrolizumab and cART) (N=12) | Cohort 3 (Pembrolizumab and cART) (N=12) | Cohort 4 (Pembrolizumab and cART) (N=24) | Total (N=58)
Anemia (Blood and lymphatic system disorders) | 5 | 10 | 7 | 11 | 33
Sinus tachycardia (Cardiac disorders) | 2 | 0 | 0 | 1 | 3
Hypothyroidism (Endocrine disorders) | 2 | 4 | 2 | 0 | 8
Blurred vision (Eye disorders) | 0 | 1 | 2 | 4 | 7
Dry eye (Eye disorders) | 0 | 1 | 0 | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 4 | 1 | 2 | 11
Bloating (Gastrointestinal disorders) | 3 | 0 | 0 | 4 | 7
Constipation (Gastrointestinal disorders) | 5 | 3 | 4 | 5 | 17
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 3 | 3 | 8
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 5 | 6
Nausea (Gastrointestinal disorders) | 5 | 2 | 5 | 7 | 19
Vomiting (Gastrointestinal disorders) | 0 | 4 | 4 | 3 | 11
Chills (General disorders) | 1 | 1 | 1 | 0 | 3
Edema limbs (Blood and lymphatic system disorders) | 5 | 1 | 0 | 2 | 8
Fatigue (General disorders) | 6 | 9 | 6 | 9 | 30
Fever (General disorders) | 2 | 2 | 1 | 3 | 8
Night sweats (General disorders) | 0 | 1 | 1 | 2 | 4
Non-cardiac chest pain (General disorders) | 1 | 1 | 1 | 1 | 4
Pain (General disorders) | 2 | 2 | 1 | 5 | 13
Upper respiratory infection (Infections and infestations) | 0 | 4 | 0 | 1 | 5
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 3
Alanine aminotransferase increased (Investigations) | 2 | 4 | 4 | 4 | 14
Alkaline phosphatase increased (Investigations) | 2 | 6 | 5 | 0 | 13
Aspartate aminotransferase increased (Investigations) | 3 | 4 | 4 | 7 | 18
Blood bilirubin increased (Investigations) | 2 | 2 | 1 | 4 | 9
CD4 lymphocytes decreased (Investigations) | 3 | 6 | 3 | 5 | 17
CPK increased (Investigations) | 0 | 1 | 5 | 15 | 21
Creatinine increased (Investigations) | 1 | 6 | 3 | 8 | 18
Lymphocyte count decreased (Investigations) | 6 | 9 | 3 | 10 | 28
Neutrophil count decreased (Investigations) | 2 | 4 | 0 | 6 | 12
Platelet count decreased (Investigations) | 2 | 3 | 2 | 3 | 10
Weight loss (Investigations) | 1 | 1 | 1 | 0 | 3
White blood cell decreased (Investigations) | 3 | 4 | 3 | 7 | 17
Anorexia (Metabolism and nutrition disorders) | 5 | 2 | 3 | 4 | 14
Hypercalcemia (Investigations) | 3 | 0 | 1 | 1 | 5
Hyperglycemia (Investigations) | 1 | 4 | 3 | 9 | 17
Hyperkalemia (Investigations) | 1 | 3 | 1 | 1 | 6
Hypoalbuminemia (Investigations) | 3 | 5 | 2 | 4 | 14
Hypocalcemia (Investigations) | 0 | 1 | 3 | 3 | 7
Hypokalemia (Investigations) | 3 | 1 | 2 | 6 | 12
Hypomagnesemia (Investigations) | 0 | 2 | 1 | 4 | 7
Hyponatremia (Investigations) | 4 | 6 | 4 | 12 | 26
Hypophosphatemia (Investigations) | 2 | 5 | 2 | 6 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 4 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4 | 4 | 12
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 2 | 5
Headache (Nervous system disorders) | 1 | 2 | 3 | 6 | 12
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 2 | 1 | 5
Anxiety (Psychiatric disorders) | 2 | 3 | 2 | 1 | 8
Depression (Psychiatric disorders) | 0 | 1 | 2 | 2 | 5
Insomnia (Psychiatric disorders) | 3 | 1 | 2 | 1 | 7
Hematuria (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 3
Proteinurea (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 2 | 4 | 11
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 2 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2 | 1 | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 1 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 2 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 4 | 3 | 10
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 2 | 4 | 4 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/66/NCT02595866/Prot_SAP_000.pdf